CLINICAL TRIAL: NCT03503279
Title: A Prospective, Randomized, Single Center Study to Compare Endotracheal Tube Placement Using McGrath MAC® Video Laryngoscope Versus Macintosh Laryngoscope in Bariatric Surgery Patients
Brief Title: Endotracheal Tube Placement Using McGrath MAC® Video Laryngoscope Versus Macintosh Laryngoscope
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started. PI left our institution and no other PI was identified
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Juan Fiorda, Post Doctoral Scholar, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017H0236
Record Dates: First submitted 2018-03-22; First posted 2018-04-19 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Macintosh Laryngoscope (No Intervention)
- McGrath MAC® Video Laryngoscope (Active Comparator)
  Interventions: Device: McGrath MAC® Video Laryngoscope

INTERVENTIONS:
Device: McGrath MAC® Video Laryngoscope — McGrath MAC® Video Laryngoscope have been developed to secure the airway and improve the management of difficult intubation. McGrath MAC® is a self-contained VL with a single-use blade; its structure is similar to the ML, but without the channel that guides the tube and a mounted LCD screen on the handle that is connected to a miniature camera with a light source at the tip of the blade, allowing the clinicians to directly observe surrounding anatomical airway structures during a tracheal intubation
  Arms: McGrath MAC® Video Laryngoscope

SUMMARY:
This study aims...

* To assess the difference in intubation difficulty scale (IDS) score following ETT placement using McGrath MAC® video laryngoscope versus conventional intubation with Macintosh laryngoscope for bariatric surgery patients
* To assess the difference in hemodynamic stimulation (airway manipulation) events in both groups
* To assess the overall difference of the duration (seconds) of ETT placement between both groups
* To assess the difference of the duration (seconds) of ETT placement during every attempt (maximum of three attempts) between both groups.
* To assess the difference of STOP BANG score between both groups
* To assess the number of intubation attempts between both groups

DETAILED DESCRIPTION:
The failure to place properly an endotracheal tube (ETT) and to secure the airway is still significantly impacting morbidity and mortality in surgical and critical care settings. In addition, no assertive predictor factor will foresee the presence of difficult airway, most of them being acknowledged after anesthesia induction. The incidence of difficult intubation reported in different studies varies from 0.1% to 13%.

The gold standard device to place an ETT that has been used since 1943 is the Macintosh laryngoscope (ML). However, in contemplation of addressing these challenging factors related to endotracheal intubation failure, modern airway devices technology has been developed in order to improve orotracheal visualization, reduce orotracehal manipulation and ensure airway patency.

As part of these novel devices, several video laryngoscopies (VL) have s been developed to secure the airway and improve the management of difficult intubation. Difficult Airway Society (DAS) guidelines recognizes the usefulness of VL in difficult intubation by providing an improved view of the airway to clinicians and directly observe/report the effects of laryngeal manipulation.

Among several VL introduced recently, a McGrath MAC® VL was announced in 2012. McGrath MAC® is a self-contained VL with a single-use blade; its structure is similar to the ML, but without the channel that guides the tube and a mounted LCD screen on the handle that is connected to a miniature camera with a light source at the tip of the blade, allowing the clinicians to directly observe surrounding anatomical airway structures during a tracheal intubation. These features have shown a better glottis visualization and to be supportive during tracheal intubation of difficult airways.

The McGrath MAC® VL and ML are standard of care devices used according to anesthesia care providers' criteria at our institution.

A single-center, prospective, randomized, double arm study, will be conducted in order to test the following hypothesis:

Reduced manipulation of the airway using McGrath MAC® VL will lead to less hemodynamic stimulation events following intubation when compared to ML.

The non-disposable portion of the McGrath MAC® VL (upper mounted reusable video camera and the optic guide) will be cleaned between usages in accordance to manufacture catalogue and institutional policy (using disinfectants such as CIDEXTM OPA, a 0.08% paracetic acid solution or disinfecting wipes).

ELIGIBILITY:
2.2. Inclusion Criteria

1. Patients (male or female) admitted for elective bariatric surgery under general anesthesia with orotracheal intubation
2. Age > 18 years old
3. American Society of Anesthesiologists (ASA) score 1-3
4. Patients capable of consenting in English language

2.3. Exclusion Criteria

1. Potential or history of difficult airway (see pages 11 and 12)
2. Past medical history of confirmed uncontrolled gastrointestinal diseases including delayed gastric emptying, dysphagia, or other gastrointestinal motility disorders that according to the investigator will not qualify for the study
3. Patients with uncontrolled metabolic disorders (e.g., diabetes mellitus, chronic kidney disease) or conditions that according to the investigator will not qualify for the study
4. Pregnant women
5. Prisoners
6. Surgery requiring patient positioning other than supine
7. Other mental, physical, and medical conditions where subject participation is inadvisable according to the investigator judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-02-02 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in intubation difficulty scale (IDS) score following ETT placement using McGrath MAC® video laryngoscope versus conventional intubation with Macintosh laryngoscope for bariatric surgery patients | Through study completion, on average of 1 week
  The Intubation Difficulty Scale (IDS) is a mixture of subjective and objective conditions that allows a qualitative and quantitative methodology to the progressive nature of the difficulty of intubation (easy=0, slightly difficult= 0<IDS≤5, moderate to major difficult= 5<IDS, impossible intubation= ∞). It could be used to asses intubating conditions and methods with the objective of determining the relative values predictive factors of intubation difficulty and of the techniques used to decrease such difficulties. It has seven parameters that are scored after an intubation: # of intubation attempts; # of alternative techniques used; a modified Cormack grade for glottic visualization; subjective impression of the lifting force needed during laryngoscopy; the need for external laryngeal pressure to optimize glottic exposure; and the position of the vocal cords.

SECONDARY OUTCOMES:
Difference in hemodynamic stimulation (airway manipulation) events in both groupsmanipulation in both groups | within 5 minutes after orotracheal intubation
  Hemodynamic events are defined as:
  * Significant variation in heart rate (HR) (defined as an increase/ decrease in HR greater than 20% of the baseline HR levels during airway management, within 5 minutes after orotracheal intubation) and,
  * Significant variations in mean blood pressure (MBP) (defined as an increase/ decrease in MBP greater than 20% of the baseline MBP levels during airway management, within 5 minutes after orotracheal intubation).
Overall difference of the duration (seconds) of ETT placement between both groups | The length of time between the date and time when the start of endotracheal tube descent maneuver until the date and time when the tube is considered well positioned in the trachea, assessed up to 10 minutes
  • The duration of intubation is defined as the time taken from the insertion of the blade beyond the incisors until the verification of the presence of three consecutive normal capnography wave forms.
Difference of the duration (seconds) of ETT placement during every attempt (maximum of three attempts) between both groups. | Procedure (The duration of intubation is defined as the time taken from the insertion of the blade beyond the incisors until the verification of the presence of three consecutive normal capnography wave forms.)
  Difference of the duration (seconds) of ETT placement
Difference of STOP BANG score between both groups | Baseline (Preoperative)
  Do you SNORE loudly (louder than talking or loud enough to be heard through closed doors)? Yes = 1 No = 0 Do you often feel TIRED, fatigued, or sleepy during daytime? Yes = 1 No = 0 Has anyone OBSERVED you stop breathing during your sleep? Yes = 1 No = 0 Do you have or are you being treated for high blood PRESSURE? Yes = 1 No = 0
  BANG BMI more than 35kg/m2? Yes = 1 No = 0 AGE over 50 years old? Yes = 1 No = 0 NECK circumference > 16 inches (40cm)? Yes = 1 No = 0 GENDER: Male? Yes = 1 No = 0
Number of intubation attempts between both groups | Procedure (Time starting at first attempt to successful attempt)
  Number of intubation attempts

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Bergese, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States